CLINICAL TRIAL: NCT00286442
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of SYR110322 (SYR-322) When Used in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Alogliptin Combined With Metformin in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322-MET-008; 2005-004668-22 (EudraCT Number); U1111-1113-8393 (Registry Identifier: WHO)
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — alogliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin and metformin
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin and metformin
- Metformin (Placebo Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Alogliptin and metformin — Alogliptin 12.5 mg, tablets, orally, once daily and metformin for up to 26 weeks.
  Other Names: alogliptin; SYR110322; Glucophage; SYR-322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin and metformin — Alogliptin 25 mg, tablets, orally, once daily and metformin for up to 26 weeks.
  Other Names: alogliptin; SYR110322; Glucophage; SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Metformin — Alogliptin placebo-matching tablets, orally, once daily and metformin for up to 26 weeks.
  Other Names: Glucophage
  Arms: Metformin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of alogliptin, once daily (QD), combined with metformin in adults with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
There are approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, of which 90% to 95% are type 2. The prevalence of type 2 diabetes varies among racial and ethnic populations and has been shown to correlate with age, obesity, family history, history of gestational diabetes, and physical inactivity. Over the next decade, a marked increase in the number of adults with diabetes mellitus is expected.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of dipeptidyl peptidase IV will improve glycemic (glucose) control in patients with type 2 diabetes.

The aim of the current study is to evaluate the effectiveness of alogliptin in combination with metformin in individually who are inadequately controlled on metformin alone.

Individuals who participate in this study will be required to commit to a screening visit and up to 14 additional visits at the study center. Study participation is anticipated to be about 34 weeks (or 8.5 months).

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of type 2 diabetes mellitus currently treated with metformin alone but, experiencing inadequate glycemic control. The participant should have received the metformin monotherapy for at least the 3 months prior to Screening; and must have a stable dose of greater than or equal to 1500 mg metformin for at least 8 weeks prior to randomization. Participants with a maximum tolerated dose that is documented to be less than 1500 mg of metformin may also be enrolled if this dose has been stable for 8 weeks prior to randomization.
* No treatment with antidiabetic agents other than metformin within the 3 months prior to Screening. (Exception: if a participant has received other antidiabetic therapy for less than 7 days within the 3 months prior to Screening.)
* Body mass index greater than or equal to 23 kg/m2 and less than or equal to 45 kg/m2
* Fasting C-peptide concentration greater than or equal to 0.8 ng per mL. (If this screening criterion is not met, the participant still qualifies if C-peptide is greater than or equal to 1.5 ng per mL after a challenge test.
* Glycosylated hemoglobin concentration between 7.0% and 10.0%, inclusive
* If regular use of other, non-excluded medications, must be on a stable dose for at least the 4 weeks prior to Screening. However, as needed use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
* Systolic blood pressure less than or equal to 180 mm Hg and diastolic pressure less than or equal to 110 mm Hg
* Hemoglobin greater than or equal to 12 g per dL for males and greater than or equal to 10 g per dL for females
* Alanine aminotransferase less than or equal to 3 time the upper limit of normal
* Serum creatinine less than1.5 mg per dL for males and less than 1.4 mg per dL for females
* Thyroid-stimulating hormone level less than or equal to the upper limit of the normal range and the participant is clinically euthyroid.
* Neither pregnant nor lactating.
* Female participants of childbearing potential must be practicing adequate contraception. Adequate contraception must be practiced for the duration of participation in the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor
* No major illness or debility that in the investigator's opinion prohibits the participant from completing the study
* Able and willing to provide written informed consent Exclusion Criteria
* Urine albumin to creatinine ratio of greater than 1000 μg per mg at Screening. If elevated, the participant may be rescreened within 1 week.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening. (A history of treated cervical intraepithelial neoplasia I or cervical intraepithelial neoplasia II is allowed.)
* History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening
* History of treated diabetic gastric paresis
* New York Heart Association Class III or IV heart failure regardless of therapy. Currently treated participants who are stable at Class I or II are candidates for the study.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus
* History of a psychiatric disorder that will affect the participant's ability to participate in the study
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors
* History of alcohol or substance abuse within the 2 years prior to Screening
* Receipt of any investigational drug within the 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within the 3 months prior to Screening
* Prior treatment in an investigational study of alogliptin
* Excluded Medications:

  * Treatment with antidiabetic agents other than study drug or metformin is not allowed within the 3 months prior to Screening and through the completion of the end-of treatment/early termination procedures.
  * Treatment with weight-loss drugs, any investigational antidiabetics, or oral or systemically injected glucocorticoids is not allowed from 3 months prior to randomization through the completion of the end-of-treatment/early termination procedures. Inhaled corticosteroids are allowed.
  * Participants must be instructed not to take any medications, including over-the-counter products, without first consulting with the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (56):
- United States (40):
  - Phoenix, Arizona
  - Anaheim, California
  - Artesia, California
  - Fresno, California
  - Los Angeles, California
  - Mission Viejo, California
  - Northridge, California
  - Orange, California
  - San Diego, California
  - Walnut Creek, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Cocoa Beach, Florida
  - Longwood, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Saint Cloud, Florida
  - Honolulu, Hawaii
  - Avon, Indiana
  - Elkhart, Indiana
  - Evansville, Indiana
  - St Louis, Missouri
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Burlington, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Pinehurst, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Medford, Oregon
  - Lansdale, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Corpus Christi, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Texarkana, Texas
  - Burlington, Vermont
- Multiple Cities, Argentina
- Multiple Cities, Australia
- Multiple Cities, Brazil
- Multiple Cities, Chile
- Multiple Cities, Czechia
- Multiple Cities, Germany
- Multiple Cities, Guatemala
- Multiple Cities, Hungary
- Multiple Cities, India
- Multiple Cities, Mexico
- Multiple Cities, Netherlands
- Multiple Cities, New Zealand
- Multiple Cities, Peru
- Multiple Cities, Poland
- Multiple Cities, South Africa
- Multiple Cities, United Kingdom

REFERENCES:
- [Result] Nauck MA, Ellis GC, Fleck PR, Wilson CA, Mekki Q; Alogliptin Study 008 Group. Efficacy and safety of adding the dipeptidyl peptidase-4 inhibitor alogliptin to metformin therapy in patients with type 2 diabetes inadequately controlled with metformin monotherapy: a multicentre, randomised, double-blind, placebo-controlled study. Int J Clin Pract. 2009 Jan;63(1):46-55. doi: 10.1111/j.1742-1241.2008.01933.x. PMID 19125992
- [Result] Pratley RE, McCall T, Fleck PR, Wilson CA, Mekki Q. Alogliptin use in elderly people: a pooled analysis from phase 2 and 3 studies. J Am Geriatr Soc. 2009 Nov;57(11):2011-9. doi: 10.1111/j.1532-5415.2009.02484.x. Epub 2009 Sep 30. PMID 19793357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 115 investigative sites in Australia, Brazil, Chile, Germany, Guatemala, Hungary, India, Mexico, New Zealand, The Netherlands, Poland, South Africa, Spain, and the United States from 10 March 2006 to 12 June 2007.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus who were inadequately controlled while receiving a stable dose of metformin monotherapy were enrolled in one of 3, once-daily (QD) treatment groups.
Groups:
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily and metformin for up to 26 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily and metformin for up to 26 weeks.
- Placebo: Alogliptin placebo-matching tablets, orally, once daily and metformin for up to 26 weeks.
Period: Overall Study
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Started | 213 | 210 | 104
Completed | 176 | 165 | 72
Not Completed | 37 | 45 | 32
Not completed — Hyperglycemic Rescue | 19 | 17 | 25
Not completed — Adverse Event | 7 | 6 | 1
Not completed — Protocol Violation | 2 | 4 | 2
Not completed — Lost to Follow-up | 5 | 2 | 1
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Administrative Error | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 14 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo | Total
Number analyzed (Participants) | 213 | 210 | 104 | 527
Age, Customized [Number; unit: participants]
  <65 years | 173 | 179 | 83 | 435
  ≥65 years | 40 | 31 | 21 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 96 | 54 | 262
  Male | 101 | 114 | 50 | 265

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26.
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 26 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had an HbA1c measurement at baseline and at Week 26.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 203 | 103
percentage of Glycosylated Hemoglobin | -0.61 (0.053) | -0.59 (0.054) | -0.10 (0.076)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Null Hypothesis: No difference between treatment and placebo arms in change from baseline in glycosylated hemoglobin at wk 26. Sample size calculated based on normally distributed means. For comparison of either dose vs. placebo (2-sample t-test), study sample size >=500 participants had 95% power to detect a treatment difference as small as 0.4% in the supportive per protocol analysis set assuming SD=0.8%, 2-sided >0.05 significance level and >=80% of participants meeting per protocol criteria; Test type: Superiority or Other; p < 0.001, ANCOVA — A step-down strategy was used for the primary analysis. First, the 25mg dose was compared to placebo at the 2-sided 0.05 significance level. The 12.5 mg dose was compared to placebo only if the comparison of the 25mg dose to placebo was significant; Analysis of covariance (ANCOVA) with treatment and geographic region as class variables and baseline metformin dose and baseline HbA1c as covariates; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.68 to -0.32] — Negative mean treatment difference indicates larger decrease from baseline (more negative change from baseline) in the alogliptin arm compared to the placebo arm
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Null Hypothesis: No difference between treatment and placebo arms in change from baseline in glycosylated hemoglobin at week 26. Sample size calculated based on normally distributed means. For comparison of either dose vs. placebo (2-sample t-test), study sample size >=500 participants had 95% power to detect a treatment difference as small as 0.4% in the per protocol analysis set assuming SD=0.8%, 2-sided test at 0.05 significance level and >=80% of participants meeting per protocol criteria; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA on change from baseline with treatment and geographic region as class variables and baseline metformin dose and baseline HbA1c as covariates; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.67 to -0.30] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had an HbA1c measurement at baseline and at Week 4. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 188 | 187 | 91
percentage of Glycosylated Hemoglobin | -0.36 (0.031) | -0.40 (0.031) | -0.10 (0.044)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.37 to -0.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.40 to -0.19] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had an HbA1c measurement at baseline and at Week 8.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 201 | 103
percentage of Glycosylated Hemoglobin | -0.59 (0.041) | -0.59 (0.042) | -0.21 (0.058)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.52 to -0.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.52 to -0.24] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had an HbA1c measurement at baseline and at Week 12.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 203 | 103
percentage of Glycosylated Hemoglobin | -0.66 (0.047) | -0.66 (0.048) | -0.16 (0.067)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.66 to -0.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.66 to -0.34] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had an HbA1c measurement at baseline and at Week 16.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 203 | 103
percentage of Glycosylated Hemoglobin | -0.66 (0.050) | -0.64 (0.051) | -0.13 (0.072)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.70 to -0.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.69 to -0.34] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had an HbA1c measurement at baseline and at Week 20.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 203 | 103
percentage of Glycosylated Hemoglobin | -0.63 (0.051) | -0.63 (0.052) | -0.12 (0.073)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.69 to -0.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.69 to -0.34] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 1).
Description: The change between the value of fasting plasma glucose collected at final visit or week 1 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 1.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 1.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 193 | 186 | 98
mg/dL | -14.3 (2.05) | -12.5 (2.09) | -0.6 (2.88)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates. Missing data imputed with LOCF; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-20.7 to -6.8] — Negative mean treatment difference indicates larger decrease from baseline (more negative change from baseline) in the alogliptin arm compared to the metformin arm
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -11.9, 95% CI 2-sided [-18.9 to -4.9] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 2.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 2.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 208 | 199 | 104
mg/dL | -17.4 (2.11) | -17.6 (2.16) | -0.7 (2.99)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-23.9 to -9.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -16.8, 95% CI 2-sided [-24.1 to -9.6] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 2. Missing data imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 204 | 104
mg/dL | -18.4 (1.98) | -18.1 (2.01) | -0.6 (2.82)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -17.8, 95% CI 2-sided [-24.6 to -11.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -17.5, 95% CI 2-sided [-24.3 to -10.6] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 8. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 204 | 104
mg/dL | -19.6 (2.30) | -17.2 (2.34) | 0.4 (3.29)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -20.1, 95% CI 2-sided [-28.0 to -12.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -17.6, 95% CI 2-sided [-25.6 to -9.7] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 12. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 204 | 104
mg/dL | -16.9 (2.44) | -16.8 (2.47) | 0.3 (3.48)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -17.2, 95% CI 2-sided [-25.6 to -8.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -17.0, 95% CI 2-sided [-25.4 to -8.6] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 16).
Description: The change between the value of fasting plasma glucose collected at week 16 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 16.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 16. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 204 | 104
mg/dL | -17.8 (2.43) | -15.4 (2.46) | 1.3 (3.46)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -19.1, 95% CI 2-sided [-27.4 to -10.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-25.0 to -8.3] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 20).
Description: The change between the value of fasting plasma glucose collected at week 20 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 20. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 204 | 104
mg/dL | -18.1 (2.53) | -15.6 (2.57) | -0.1 (3.61)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -18.1, 95% CI 2-sided [-26.7 to -9.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -15.5, 95% CI 2-sided [-24.2 to -6.8] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 26).
Description: The change between the value of fasting plasma glucose collected at week 26 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 204 | 104
mg/dL | -18.7 (2.49) | -17.4 (2.53) | 0.0 (3.55)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -18.7, 95% CI 2-sided [-27.3 to -10.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -17.4, 95% CI 2-sided [-25.9 to -8.8] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Number of Participants With Marked Hyperglycemia (Fasting Plasma Glucose ≥ 200 mg Per dL).
Description: The number of participants with a fasting plasma glucose value greater than or equal to 200 mg per dL during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had at least 1 fasting plasma glucose measurement after baseline.
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 206 | 104
participants | 61 | 65 | 53
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — no multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 0.372, 95% CI 2-sided [0.213 to 0.650] — Odd's Ratio (OR) is alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 0.405, 95% CI 2-sided [0.231 to 0.708] — Odd's Ratio (OR) is alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

16. Secondary Outcome: Number of Participants Requiring Rescue.
Description: The number of participants requiring rescue for failing to achieve pre-specified glycemic targets during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who completed at least 1 study visit after baseline.
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 211 | 207 | 104
participants | 19 | 17 | 25
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Logistic — no multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 0.302, 95% CI 2-sided [0.143 to 0.635] — Odd's Ratio (OR) is alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 0.236, 95% CI 2-sided [0.109 to 0.510] — Odd's Ratio (OR) is alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

17. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 4).
Description: The change between the value of fasting proinsulin collected at week 4 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a fasting plasma glucose measurement at baseline and at Week 4. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 178 | 174 | 90
pmol/L | -1.9 (1.76) | -5.0 (1.77) | -0.5 (2.47)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.634, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-7.4 to 4.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.136, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-10.5 to 1.4] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 8).
Description: The change between the value of fasting proinsulin collected at week 8 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a proinsulin measurement at baseline and at Week 8. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 201 | 189 | 100
pmol/L | -2.9 (1.30) | -5.0 (1.34) | -0.4 (1.85)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.274, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-6.9 to 2.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.046, ANCOVA — No multiplicity adjustments; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-9.1 to -0.1] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 12).
Description: The change between the value of fasting proinsulin collected at week 12 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a proinsulin measurement at baseline and at Week 12. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 201 | 191 | 100
pmol/L | -2.6 (1.76) | -2.7 (1.8) | -1.3 (2.49)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.655, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-7.4 to 4.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.645, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline FPG as covariates; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-7.4 to 4.6] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 16).
Description: The change between the value of fasting proinsulin collected at week 16 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a proinsulin measurement at baseline and at Week 16. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 201 | 191 | 100
pmol/L | -1.4 (1.60) | -2.7 (1.64) | -0.5 (2.26)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.748, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-6.3 to 4.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.432, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-7.7 to 3.3] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 20).
Description: The change between the value of fasting proinsulin collected at week 20 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a proinsulin measurement at baseline and at Week 20. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 201 | 191 | 100
pmol/L | -4.2 (1.62) | -1.1 (1.66) | -2.0 (2.29)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.427, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-7.8 to 3.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.746, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-4.6 to 6.5] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 26).
Description: The change between the value of fasting proinsulin collected at week 26 or final visit and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a PROINSULIN measurement at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 201 | 191 | 100
pmol/L | -2.1 (1.80) | -1.6 (1.84) | -3.2 (2.54)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.727, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-5.0 to 7.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 1.6, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin as covariates; Mean Difference (Final Values) = 0.601, 95% CI 2-sided [-4.5 to 7.8] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Change From Baseline in Insulin (Week 4).
Description: The change between the value of insulin collected at week 4 and insulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had an insulin measurement at baseline and at Week 4. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 177 | 170 | 89
mcIU/mL | 1.11 (0.684) | 0.52 (0.695) | -1.07 (0.965)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.066, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 2.19, 95% CI 2-sided [-0.15 to 4.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.180, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [-0.74 to 3.93] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Change From Baseline in Insulin (Week 8).
Description: The change between the value of insulin collected at week 8 and insulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a Insulin measurement at baseline and at Week 8. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 186 | 99
mcIU/mL | 2.50 (1.416) | 0.18 (1.466) | 2.68 (2.015)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.944, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-5.02 to 4.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.316, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-7.40 to 2.40] — [estimate comment as in outcome 1, analysis 1]

25. Secondary Outcome: Change From Baseline in Insulin (Week 12).
Description: The change between the value of insulin collected at week 12 and insulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a Insulin measurement at baseline and at Week 12. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
mcIU/mL | 1.6 (1.488) | 0.46 (1.532) | 1.92 (2.118)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.901, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-5.42 to 4.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.578, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-6.59 to 3.68] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Change From Baseline in Insulin (Week 16).
Description: The change between the value of insulin collected at week 16 and insulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a Insulin measurement at baseline and at Week 16. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
mcIU/mL | 1.27 (0.964) | 1.53 (0.993) | 0.64 (1.372)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.708, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-2.67 to 3.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.601, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-2.44 to 4.21] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Change From Baseline in Insulin (Week 20).
Description: The change between the value of insulin collected at week 20 and insulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a Insulin measurement at baseline and at Week 20. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
mcIU/mL | 0.91 (0.760) | 0.86 (0.782) | -0.21 (1.081)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.398, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-1.48 to 3.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.425, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 1.07, 95% CI 2-sided [-1.56 to 3.69] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Change From Baseline in Insulin (Week 26).
Description: The change between the value of insulin collected at week 26 and insulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had a Insulin measurement at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
mcIU/mL | 0.63 (0.690) | -0.01 (0.710) | -2.23 (0.981)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 2.87, 95% CI 2-sided [0.50 to 5.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.067, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline insulin as covariates; Mean Difference (Final Values) = 2.22, 95% CI 2-sided [-0.15 to 4.60] — [estimate comment as in outcome 1, analysis 1]

29. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 4).
Description: The change between the ratio value of proinsulin and insulin collected at week 4 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had insulin and proinsulin measurements at baseline and at Week 4. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 177 | 170 | 89
ratio | -0.045 (0.0082) | -0.056 (0.0083) | -0.008 (0.0115)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline proinsulin/insulin ratio as covariates; Mean Difference (Final Values) = -0.036, 95% CI 2-sided [-0.064 to -0.009] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.047, 95% CI 2-sided [-0.075 to -0.019] — [estimate comment as in outcome 1, analysis 1]

30. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 8).
Description: The change between the ratio value of proinsulin and insulin collected at week 8 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had insulin and proinsulin measurements at baseline and at Week 8. Missing data are imputed using last observation carried forward (LOCF.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 186 | 99
ratio | -0.055 (0.0073) | -0.046 (0.0075) | -0.009 (0.0103)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.045, 95% CI 2-sided [-0.070 to -0.021] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.037, 95% CI 2-sided [-0.062 to -0.012] — [estimate comment as in outcome 1, analysis 1]

31. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 12).
Description: The change between the ratio value of proinsulin and insulin collected at week 12 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had insulin and proinsulin measurements at baseline and at Week 12. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
ratio | -0.044 (0.0083) | -0.042 (0.0085) | -0.005 (0.0118)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.039, 95% CI 2-sided [-0.068 to -0.011] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.037, 95% CI 2-sided [-0.066 to -0.008] — [estimate comment as in outcome 1, analysis 1]

32. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 16).
Description: The change between the ratio value of proinsulin and insulin collected at week 16 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had insulin and proinsulin measurements at baseline and at Week 16. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
ratio | -0.051 (0.0082) | -0.043 (0.0085) | 0.001 (0.0117)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.052, 95% CI 2-sided [-0.080 to -0.024] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.044, 95% CI 2-sided [-0.072 to -0.015] — [estimate comment as in outcome 1, analysis 1]

33. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 20).
Description: The change between the ratio value of proinsulin and insulin collected at week 20 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had insulin and proinsulin measurements at baseline and at Week 20. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
ratio | -0.53 (0.0150) | -0.011 (0.0155) | -0.007 (0.0213)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.078, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.046, 95% CI 2-sided [-0.097 to 0.005] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.860, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.056 to 0.047] — [estimate comment as in outcome 1, analysis 1]

34. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 26).
Description: The change between the ratio value of proinsulin and insulin collected at week 26 or final visit and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had insulin and proinsulin measurements at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 200 | 188 | 99
ratio | -0.049 (0.0154) | 0.000 (0.0159) | 0.004 (0.0219)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.048, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.053, 95% CI 2-sided [-0.106 to -0.001] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.889, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.057 to 0.050] — [estimate comment as in outcome 1, analysis 1]

35. Secondary Outcome: Change From Baseline in C-peptide (Week 4).
Description: The change between the value of C-peptide collected at week 4 and C-peptide collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had C-peptide measurements at baseline and at Week 4. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 186 | 184 | 92
ng/mL | 0.222 (0.0893) | 0.190 (0.0897) | -0.114 (0.1273)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.031, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.336, 95% CI 2-sided [0.030 to 0.642] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.051, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.304, 95% CI 2-sided [-0.002 to 0.611] — [estimate comment as in outcome 1, analysis 1]

36. Secondary Outcome: Change From Baseline in C-peptide (Week 8).
Description: The change between the value of C-peptide collected at week 8 and C-peptide collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had C-peptide measurements at baseline and at Week 8. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 200 | 103
ng/mL | 0.215 (0.0864) | 0.238 (0.0884) | 0.127 (0.1236)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.563, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.088, 95% CI 2-sided [-0.209 to 0.384] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.467, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [-0.188 to 0.410] — [estimate comment as in outcome 1, analysis 1]

37. Secondary Outcome: Change From Baseline in C-peptide (Week 12).
Description: The change between the value of C-peptide collected at week 12 and C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had C-peptide measurements at baseline and at Week 12. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 202 | 103
ng/mL | 0.154 (0.0915) | 0.246 (0.0932) | -0.033 (0.1309)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.243, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.187, 95% CI 2-sided [-0.127 to 0.501] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.083, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.279, 95% CI 2-sided [-0.037 to 0.595] — [estimate comment as in outcome 1, analysis 1]

38. Secondary Outcome: Change From Baseline in C-peptide (Week 16).
Description: The change between the value of C-peptide collected at week 16 and C-peptide collected at baseline.
Time Frame: Baseline and Week 16.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had C-peptide measurements at baseline and at Week 16. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 202 | 103
ng/mL | 0.138 (0.0894) | 0.250 (0.0910) | -0.018 (0.1280)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.321, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.155, 95% CI 2-sided [-0.152 to 0.463] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.089, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.268, 95% CI 2-sided [-0.041 to 0.577] — [estimate comment as in outcome 1, analysis 1]

39. Secondary Outcome: Change From Baseline in C-peptide (Week 20).
Description: The change between the value of C-peptide collected at week 20 and C-peptide collected at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had C-peptide measurements at baseline and at Week 20. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 202 | 103
ng/mL | 0.007 (0.0803) | 0.054 (0.0818) | -0.137 (0.1149)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.305, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [-0.132 to 0.420] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.177, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.191, 95% CI 2-sided [-0.086 to 0.468] — [estimate comment as in outcome 1, analysis 1]

40. Secondary Outcome: Change From Baseline in C-peptide (Week 26).
Description: The change between the value of C-peptide collected at week 26 or final visit and C-peptide collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had C-peptide measurements at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 210 | 202 | 103
ng/mL | -0.083 (0.0833) | -0.214 (0.0848) | -0.476 (0.1192)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.394, 95% CI 2-sided [0.107 to 0.680] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.074, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline C-peptide as covariates; Mean Difference (Final Values) = 0.263, 95% CI 2-sided [-0.025 to 0.550] — [estimate comment as in outcome 1, analysis 1]

41. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 6.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 6.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 213 | 207 | 104
participants | 42 | 36 | 4
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — no multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 6.150, 95% CI 2-sided [2.117 to 17.864] — Odd's Ratio (OR) is alogliptin arm versus placebo. OR >1.0 indicates higher incidence of response compared to placebo
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 5.322, 95% CI 2-sided [1.820 to 15.564] — Odd's Ratio (OR) is alogliptin arm versus placebo. OR >1.0 indicates higher incidence of response compared to placebo

42. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.0%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 7.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 213 | 207 | 104
participants | 110 | 92 | 19
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 6.092, 95% CI 2-sided [3.271 to 11.345] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR >1.0 indicates higher incidence of response compared to placebo
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 4.451, 95% CI 2-sided [2.388 to 8.296] — [estimate comment as in outcome 42, analysis 1]

43. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 7.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 213 | 207 | 104
participants | 153 | 137 | 47
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 4.238, 95% CI 2-sided [2.327 to 7.717] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 3.293, 95% CI 2-sided [1.814 to 5.979] — [estimate comment as in outcome 42, analysis 1]

44. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 0.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 0.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 213 | 207 | 104
participants | 123 | 122 | 28
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 4.103, 95% CI 2-sided [2.428 to 6.934] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 4.314, 95% CI 2-sided [2.545 to 7.312] — [estimate comment as in outcome 42, analysis 1]

45. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 213 | 207 | 104
participants | 61 | 62 | 9
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 5.601, 95% CI 2-sided [2.554 to 12.282] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 5.793, 95% CI 2-sided [2.645 to 12.684] — [estimate comment as in outcome 42, analysis 1]

46. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 213 | 207 | 104
participants | 20 | 24 | 6
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.085, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 2.449, 95% CI 2-sided [0.883 to 6.797] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.034, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 2.958, 95% CI 2-sided [1.087 to 8.046] — [estimate comment as in outcome 42, analysis 1]

47. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 2.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 2.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 213 | 207 | 104
participants | 7 | 5 | 4
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.639, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 1.404, 95% CI 2-sided [0.340 to 5.803] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.956, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin dose and baseline HbA1c; Odds Ratio (OR) = 0.959, 95% CI 2-sided [0.218 to 4.223] — [estimate comment as in outcome 42, analysis 1]

48. Secondary Outcome: Change From Baseline in Body Weight (Week 8).
Description: The change between Body Weight measured at week 8 and Body Weight measured at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had weight measurements at baseline and at Week 8. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 198 | 193 | 102
kg | -0.30 (0.134) | -0.53 (0.135) | -0.12 (0.186)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.439, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.63 to 0.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.075, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.86 to 0.04] — [estimate comment as in outcome 1, analysis 1]

49. Secondary Outcome: Change From Baseline in Body Weight (Week 12).
Description: The change between Body Weight measured at week 12 and Body Weight measured at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had weight measurements at baseline and at Week 12. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 205 | 198 | 103
kg | -0.28 (0.161) | -0.64 (0.164) | -0.57 (0.227)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.305, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.26 to 0.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.788, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.63 to 0.47] — [estimate comment as in outcome 1, analysis 1]

50. Secondary Outcome: Change From Baseline in Body Weight (Week 20).
Description: The change between Body Weight measured at week 20 and Body Weight measured at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had weight measurements at baseline and at Week 20. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 205 | 198 | 103
kg | -0.38 (0.178) | -0.58 (0.182) | -0.40 (0.252)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.930, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.58 to 0.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.559, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.79 to 0.43] — [estimate comment as in outcome 1, analysis 1]

51. Secondary Outcome: Change From Baseline in Body Weight (Week 26).
Description: The change between Body Weight measured at week 26 or final visit and Body Weight measured at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least 1 dose of study drug (Full Analysis Set), and who had weight measurements at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Number analyzed (Participants) | 206 | 198 | 103
kg | -0.39 (0.194) | -0.67 (0.198) | -0.39 (0.274)
Statistical Analysis 1: Comparison: Alogliptin 12.5 mg QD vs Placebo; Test type: Superiority or Other; p = 0.996, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.66 to 0.66] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin 25 mg QD vs Placebo; Test type: Superiority or Other; p = 0.407, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; baseline metformin dose and baseline weight as covariates; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.94 to 0.38] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Placebo
Serious Adverse Events (participants affected / at risk) | 6/213 | 8/207 | 4/104
Other Adverse Events (participants affected / at risk) | 62/213 | 41/207 | 37/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD (N=213) | Alogliptin 25 mg QD (N=207) | Placebo (N=104)
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-secretory adenoma of the pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD (N=213) | Alogliptin 25 mg QD (N=207) | Placebo (N=104)
Upper respiratory tract infection (Infections and infestations) | 10 | 5 | 7
Urinary tract infection (Infections and infestations) | 14 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 7 | 6
Nasopharyngitis (Infections and infestations) | 12 | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5
Hypertension (Vascular disorders) | 4 | 6 | 5
Sinusitis (Infections and infestations) | 5 | 4 | 5
Bronchitis (Infections and infestations) | 9 | 6 | 2
Pain in extremity (General disorders) | 5 | 3 | 4
Headache (Nervous system disorders) | 8 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.